CLINICAL TRIAL: NCT01166932
Title: COMPARISON OF CLINICAL EFFICACY OF COMBINATION Amoxycillin Plus Clavulanic Acid and Oxacillin Plus Ceftriaxone for HOSPITAL TREATMENT OF COMMUNITY Acquired PNEUMONIA IN CHILDREN : A Randomized Clinical Study
Brief Title: Comparison Between Amoxycillin/Clavulanic Acid and Oxacillin/Ceftriaxone for Community Acquired-pneumonia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Responsible Party: Jose Roberto Fioretto, UNESP HC FM Botucatu Unesp
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: upeclin/HC/FMB-Unesp-44
Record Dates: First submitted 2010-05-11; First posted 2010-07-21 (Estimated); Last update posted 2010-11-01 (Estimated); Status verified 2010-10

CONDITIONS: Community-Acquired Pneumonia
Keywords: pneumonia; children; antibiotics
MeSH Terms: conditions — Community-Acquired Pneumonia; Pneumonia | interventions — Amoxicillin-Potassium Clavulanate Combination; Ceftriaxone; Oxacillin

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- amoxicillin/clavulanic acid (Active Comparator): patients who received amoxicillin/clavulanic acid
  Interventions: Drug: Amoxycillin/clavulanic acid
- ceftriaxone/oxacillin (Active Comparator)
  Interventions: Drug: ceftriaxone/oxacillin

INTERVENTIONS:
Drug: Amoxycillin/clavulanic acid — 100mg/Kg/day/10 days.
  Arms: amoxicillin/clavulanic acid
Drug: ceftriaxone/oxacillin — 75 mg/Kg/day/10 days.
  Arms: ceftriaxone/oxacillin

SUMMARY:
Objective: To compare the clinical effectiveness and hospital costs, the initial empirical treatment, Oxacillin / Ceftriaxone and Amoxicillin / Clavulanate in children with Community Acquired Pneumonia (CAP) severe.

Methods: Clinical prospective randomized study in children aged two months to five years of age with a diagnosis of severe CAP, according to criteria of World Health Organization (WHO), admitted to the Pediatrics Ward of the Hospital of the Medical School of Botucatu- UNESP. We excluded children with comorbid disorders (primary and secondary immunodeficiency) with acute or chronic kidney disease, referred patients receiving antibiotics proposal and history of allergy to antibiotics proposed. We included 104 children who were randomized into two groups to receive: Oxacillin / Ceftriaxone IV (GCO, n = 48) and Amoxicillin / Clavulanate IV (GAA, n = 56). Patients of the GAA, after clinical improvement, has been receiving the same oral antibiotic, and maintaining clinical stability, were discharged from hospital, the GOC received any IV treatment. The outcomes analyzed were time to clinical improvement (fever and tachypnea), duration of oxygen therapy, hospitalization time, need to expand the antimicrobial spectrum progression to pleural effusion / empyema (DP / E) and hospital costs. Treatment failure was determined by the need to expand the antimicrobial spectrum after 48 hours of hospitalization.

DETAILED DESCRIPTION:
eligibility: Children aged two months to five years with diagnosis of severe community acquired pneumonia, requiring hospitalization.

Outcomes measures: time to clinical improvement (respiratory rate and fever), duration of oxygen therapy, length of stay in the Division of Pediatrics, evolution with clinical complications, need for broadening the spectrum antimicrobials.

ELIGIBILITY:
Inclusion Criteria:

* children aged from 2 months to 5 years
* children diagnosed with severe community-acquired pneumonia, who require hospitalization.

Exclusion Criteria:

* chronical diseases
* severe comorbidities
* children admitted at PICU

Ages: 2 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2005-04; Primary Completion 2007-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
length of stay at pediatric ward. | 3 years

SECONDARY OUTCOMES:
need for broadening the spectrum antimicrobials. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Cristiane F Ribeiro, MD, Principal Investigator — UNESP - Botucatu Medical School
Locations (1):
- Cristiane Franco Ribeiro, Botucatu, São Paulo, Brazil

REFERENCES:
- [Derived] Ribeiro CF, Ferrari GF, Fioretto JR. Antibiotic treatment schemes for very severe community-acquired pneumonia in children: a randomized clinical study. Rev Panam Salud Publica. 2011 Jun;29(6):444-50. PMID 21829969